CLINICAL TRIAL: NCT02686229
Title: Registry Study on Epidemiological and Biological Disease Profile as Well as Clinical Outcome in Patients With Low Grade Gliomas: The LOG-Glio-Project
Brief Title: Registry Study on Epidemiological and Biological Disease Profile as Well as Clinical Outcome in Patients With Low Grade Gliomas
Acronym: LoG-Glio
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jan Coburger, M.D., University of Ulm
Other Study IDs: LoG-Glio
Record Dates: First submitted 2016-02-04; First posted 2016-02-19 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Glioma
Keywords: Low grade glioma, registry, neurosurgery, brain tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood and tumor samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: no interventions

SUMMARY:
The LoG-Glio-Registry is based on a network of german hospitals gathering radiological, clinical, epidemiological and molecular data on all patients diagnosed with a low grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiological suspected diagnosis of a low grade glioma
* Age ≥ 18 years. There is no upper age limit.

Exclusion Criteria:

* Severe neurological or psychiatric disorder interfering with ability to give an informed consent
* No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician about study participation
* No consent for bio-banking of patient's biological specimens and performance of analyses on stored material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with radiological suspected diagnosis of a low grade glioma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5yrs
Overall survival (OS) | 15yrs

SECONDARY OUTCOMES:
Extent of tumor resection | 3yrs
  calculated based on volumetric assessement of tumor in cm³ and residual tumor in pre and postoperative MRI
Quality of life (QoL) assessed by the EORTC QLQ C-30/BN-20. (European Organisation for Research and Treatment of Cancer Quality of Life Questionaire C-30 | 5yrs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pala A, Nadji-Ohl M, Faust K, Ruckriegel S, Roder C, von der Brelie C, Forster MT, Lobel F, Schommer S, Lohr M, Renovanz M, Grubel N, Rothenbacher D, Konig R, Engelke J, Schmitz B, Wirtz CR, Ringel F, Senft C, Rohde V, Tatagiba M, Ernestus RI, Vajkoczy P, Ganslandt O, Nagel G, Coburger J. Multicentric Registry Study on Epidemiological and Biological Disease Profile as Well as Clinical Outcome in Patients with Low-Grade Gliomas: The LoG-Glio Project. J Neurol Surg A Cent Eur Neurosurg. 2020 Jan;81(1):48-57. doi: 10.1055/s-0039-1693650. Epub 2019 Sep 24. PMID 31550737